CLINICAL TRIAL: NCT01428089
Title: Suppression of Daytime and Nighttime LH Frequency by Progesterone in Early Pubertal Girls With and Without Hyperandrogenemia (JCM024)
Brief Title: Suppression of Daytime and Nighttime Luteinizing Hormone Frequency by Progesterone
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Chris McCartney, Center for Research in Reproduction, University of Virginia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 13660; P50HD028934 (NIH)
Record Dates: First submitted 2011-08-30; First posted 2011-09-02 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Polycystic Ovary Syndrome; Hyperandrogenism; Normal Puberty
Keywords: hyperandrogenemia
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hyperandrogenism | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Progesterone (Experimental): Subjects will take 5-25 mg oral micronized P (based on body weight, to achieve mean plasma P 1-2 ng/ml)
  Interventions: Drug: Progesterone
- placebo (Placebo Comparator): placebo at 1100, 1500, and 1900 h.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Progesterone — Subjects will take 5-25 mg oral micronized P (based on body weight, to achieve mean plasma P 1-2 ng/ml) or placebo at 1100, 1500, and 1900 h.
  Arms: Progesterone
Drug: Placebo — Placebo
  Arms: placebo

SUMMARY:
During childhood, the levels of certain hormones: gonadotropin-releasing hormone (GnRH), luteinizing hormone (LH), follicle-stimulating hormone (FSH), estrogen, and progesterone are very low. However, when puberty starts, GnRH and LH pulses begin to increase, but they initially do so at night only. It is unknown why GnRH and LH pulses increase at night and then decrease during the day (instead of being increased all the time). The purpose of this study is to see how quickly progesterone reduces LH pulses. The study is also meant to find out whether too much testosterone (also a hormone) in the blood causes problems with the ability of progesterone to reduce LH pulses. In this study, the investigators aim to discover whether or not giving 3 small doses of progesterone to pubertal girls will prevent the nighttime increase of LH pulses. From the information gathered in this study, the investigators may be able to learn more about how menstrual cycles are normally established in girls during puberty. Ultimately, if the investigators understand these normal processes, the investigators may be able to better understand abnormalities of puberty.

DETAILED DESCRIPTION:
Studies will be performed in early pubertal (late Tanner 1 [estradiol level > 20 pg/ml] to Tanner 3, premenarcheal) girls with and without hyperandrogenemia (HA). After a potential subject is identified by the Pediatric, Teen, or Endocrine clinics, she will come to the CRU or alternate UVA clinical unit for an outpatient screening exam. The goals and procedures of the study will be explained to the potential subjects and their custodial parents, and they will be given the opportunity to ask questions. A subject and her custodial parent(s) will be asked to sign the assent and consent forms. A physician will record a family and personal medical history and perform a physical exam. The physical exam will include height, weight, and determination of pubertal stage (Tanner scale). Since adiposity is a potential confounder in this study, measures of adiposity will be recorded. This will include measurement of waist circumference (using standard technique) to provide an estimate of abdominal adiposity. Hip circumference will also be measured. Additionally, BOD POD® will be used to measure total fat mass, fat free mass, and percent body fat. Blood tests will include CBC, Chem17, prolactin, LH, FSH, E2, P, total testosterone, SHBG, DHEA-S, 17-OHP, TSH, insulin, beta-hCG, and cytoadipokines. Bone age (simple x-ray of left hand and wrist) will be measured.

If safety labs are abnormal during screening (e.g., abnormal liver tests, abnormal TSH), subjects will be asked to return once for repeat (confirmatory) labs to exclude lab error, especially when values are only slightly abnormal. Repeat testing will generally occur within one month of the original screening lab draw. If exclusionary lab values are confirmed on such repeat testing, subjects will be excluded from participation. If the subject has a low hemoglobin (<11.5 g/dL for non-African American subjects; Hemoglobin < 11.0 g/dL for African American subjects ) at the time of screening, we will offer the option of taking oral iron supplementation at a dose of 1-2 mg/kg for 30 days. Subjects weighing ≤ 36 kg will be given 300-325 mg oral ferrous gluconate daily (containing 36 mg of elemental iron); subjects weighing >36 kg will be given 300-325 mg oral ferrous gluconate twice daily. Following the course of iron supplementation, the subject will then return to the CRU for a repeat hemoglobin, and will only be able to proceed with the study if her hemoglobin is greater than or equal to 11.0 g/dL for African American subjects or greater than or equal to 11.5 g/dL for non-African American subjects. If the subject's hemoglobin remains low after repeat testing, we will recommend that they follow up with their primary physician.

If three months have elapsed between an admission and the subject's most recent safety labs, then safety labs (CBC, chemistry and liver panel) will be obtained prior to the overnight admission (or on admission) to exclude anemia and any other exclusion criteria.

Subjects who meet all inclusion criteria will then be scheduled for an inpatient admission. They will begin taking iron supplementation for a maximum of 30 days prior to admission. Girls weighing ≤ 36 kg will take one 300-325 mg tablet oral ferrous gluconate daily (containing 36 mg elemental iron); subjects weighing >36 kg will take two 300-325 tablets oral ferrous gluconate daily (containing 36 mg elemental iron). The inpatient admission can occur at any time during this period of iron supplementation.

Inpatient Admission:

The subject will be admitted to the CRU, or alternate UVA hospital unit, at 0900-1000 h. A urine pregnancy test (HCG) will be obtained. A hemoglobin will be measured-if a CBC has not been done within the past 7 days, a fingerstick will be done to check the hemoglobin prior to insertion of the IV line. Alternatively, subjects may come to the CRU early on the day of their admission before their scheduled admission time. The study team will be responsible for scheduling this with the subject. In order to continue with the admission, girls must have a negative HCG. They must also have either a hemoglobin ≥ 11.0 g/dL for African American subjects or ≥ 11.5 g/dL for non-African American subjects. A small amount of topical lidocaine and prilocaine cream (EMLA cream) may be applied to facilitate IV line placement. An IV line will be placed in a forearm vein at ~1000-1030 h, and blood draws will begin at 1100 h.

Samples will be taken every 10 min for 20 h (i.e., from 1100 h to 0700 h the following day).

* Sample volume will be 0.75 ml every 10 minutes for later measurement of LH.
* Every 2 hours (on the hour), an additional 3.5 ml will be drawn for later measurement of FSH, T, E2, P, and cortisol.
* At 0700 h, an additional 3.5 ml will be drawn for measurement of fasting insulin, glucose, SHBG, DHEAS, IGF-1, and androstenedione.

Subjects will take 5-25 mg oral micronized P (based on body weight, to achieve mean plasma P 1-2 ng/ml) or placebo at 1100, 1500, and 1900 h.

Formal lights out will occur at 2300 h, and subjects will be encouraged to sleep at this time. Subjects will be awakened at 0700 h. No sleeping will be allowed from 1100-2300 h. During blood sampling, activity (e.g., awake, sleeping) will be recorded by the nurse every 10 minutes. Additionally, periods of sleep will be estimated using wrist actigraphy (Motionlogger Basic-L; Ambulatory Monitoring, Inc.) (42). The Motionlogger Basic-L is a watch-like device (that includes an accelerometer) that will be worn on the wrist by the research participant during the overnight admission.

Subjects will be fasting from 2100 to 0700 h. The subject will be offered meals at standard meal times the evening prior to study, but breakfast will not be served until after the 0700 h sample is obtained.

Optional Follow-Up for study participants: Subjects participating in this study will be asked to respond to a questionnaire (sent via electronic mail or US postal service) and/or phone calls at 6-12 month intervals during the subsequent three years to determine the progression of normal puberty, the onset and frequency of menses, and the development of any hirsutism. Whenever possible, we will see the patient in the CRU or alternate UVA clinical unit at these times to obtain blood for hormone analysis including fasting insulin and glucose, cortisol, SHBG, testosterone, DHEA-S, LH, FSH, estradiol and progesterone (10 cc of blood drawn with each visit); in addition to a brief physical exam to include height, weight, and Tanner stage. The follow-up portion of this study is completely optional.

ELIGIBILITY:
Inclusion Criteria:

* Female volunteers in early to mid-puberty (i.e., late Tanner I [estradiol level > 20 pg/mL], Tanner II, or Tanner III)
* Premenarcheal

Exclusion Criteria:

* Pregnancy
* Inability to comprehend what will be done during the study or why it will be done
* Hemoglobin less than 12 g/dl and hematocrit less than 36%
* Persistently abnormal sodium, potassium, or bicarbonate (i.e., confirmed on repeat)
* Persistently elevated creatinine, hepatic transaminases, or alkaline phosphatase (i.e., confirmed on repeat)
* Total bilirubin > 1.5 times upper limit of normal (i.e., confirmed on repeat)
* Significant history of cardiac or pulmonary dysfunction (e.g., known or suspected congestive heart failure; asthma requiring intermittent systemic corticosteroids; etc.)
* Untreated hypo- or hyperthyroidism, reflected by persistently abnormal thyroid-stimulating hormone (TSH) values
* Total testosterone > 200 ng/dl
* Basal (follicular) 17-hydroxyprogesterone > 200 ng/ml (in girls without a previous diagnosis of congenital adrenal hyperplasia)
* Dehydroepiandrosterone sulfate (DHEA-S) > 800 mcg/dl
* Elevation of prolactin > 2 times upper limit of normal
* Weight less than 26 kg.

Ages: 7 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2011-03-11 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Average luteinizing hormone (LH) interpulse interval and the total number of LH pulses | 1100hr to 0700 hr

SECONDARY OUTCOMES:
Hourly hormone measurements during sampling period. | 1100hr to 0700 hr
  The hourly measurements of progesterone, FSH, estrogen, and testosterone will be analyzed in a similar manner as the LH interpulse interval data.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R McCartney, MD, Principal Investigator — University of Virginia
Locations (1):
- Center for Research in Reproduction, University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
We do not have current plans to share IPD